CLINICAL TRIAL: NCT01483027
Title: A Phase III Clinical Trial Evaluating TheraSphere® in Patients With Metastatic Colorectal Carcinoma of the Liver Who Have Failed First Line Chemotherapy
Brief Title: Efficacy Evaluation of TheraSphere Following Failed First Line Chemotherapy in Metastatic Colorectal Cancer
Acronym: EPOCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS-102
Record Dates: First submitted 2011-11-24; First posted 2011-12-01 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Standard of care second-line chemotherapy plus TheraSphere
  Interventions: Device: TheraSphere
- Control group (No Intervention): Standard of care second-line chemotherapy with no added therapy

INTERVENTIONS:
Device: TheraSphere — yttrium 90 microspheres
  Arms: Treatment group

SUMMARY:
The effectiveness and safety of TheraSphere will be evaluated in patients with colorectal cancer with metastases in the liver, who are scheduled to receive second line chemotherapy. All patients receive the standard of care chemotherapy with or without the addition of TheraSphere.

ELIGIBILITY:
Inclusion Criteria

* Must be male or female, 18 years of age or older, and of any ethnic or racial group
* If primary tumor has not been resected, it must be clinically stable
* Must have colorectal cancer with unresectable metastatic disease to the liver (unresectable unilobar or bilobar disease) who have disease progression in the liver with oxaliplatin or irinotecan based first line chemotherapy
* Must be eligible to receive second-line standard-of-care chemotherapy with either 1) an oxaliplatin-based chemotherapy regimen, or 2) an irinotecan-based chemotherapy regimen
* Must have baseline efficacy images with measurable target tumors in the liver according to RECIST 1.1 using standard imaging techniques taken within 28 days prior to randomization. Images must be taken after, or at the time of completion of first line chemotherapy
* Tumor replacement <50% of total liver volume
* Current Eastern Cooperative Oncology Group (ECOG) of 0-1 through screening to first treatment on study
* Will have completed the first line chemotherapy regimen at least 14 days prior to initiation of 2nd line chemotherapy under the protocol
* Patient is willing to participate in the study and has signed the study informed consent
* Serum creatinine ≤ 2.0 mg/dL
* Serum bilirubin up to 1.2 x upper limit of normal
* Albumin ≥ 3.0 g/dL
* Must have neutrophil count >1200/mm3 (1.2x109/L)

Exclusion Criteria

* History of hepatic encephalopathy
* Contraindications to angiography and selective visceral catheterization such as bleeding diathesis or coagulopathy that is not correctable by usual therapy of hemostatic agents (eg. closure device)
* History of severe peripheral allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically
* Presentation of pulmonary insufficiency or clinically evident chronic obstructive pulmonary disease
* Cirrhosis or portal hypertension
* Prior external beam radiation treatment to the liver
* Prior intra-arterial liver directed therapy, including transcatheter arterial chemoembolization (TACE) or Y-90 microsphere therapy
* Planned treatment with biological agents within 28 days prior to receiving TheraSphere
* Planned liver directed therapy or radiation therapy
* Intervention for, or compromise of, the Ampulla of Vater
* Clinically evident ascites (trace ascites on imaging is acceptable)
* Toxicities due to prior cancer therapy that have not resolved before the initiation of study treatment, if the Investigator determines that the continuing complication will compromise the safe treatment of the patient
* Significant life-threatening extra-hepatic disease, including patients who are on dialysis, have unresolved diarrhea, have serious unresolved infections including patients who are known to be human immunodeficiency virus (HIV) positive or have acute hepatitis B virus (HBV) or hepatitis C virus (HCV)
* confirmed extra-hepatic metastases. Limited indeterminate extra-hepatic lesions in the lung and/or lymph nodes are permitted (up to 5 lesions in the lung, with each individual lesion <1 cm; any number of lymph nodes with each individual nodes <1.5 cm)
* Contraindications to the planned second line standard-of-care chemotherapy regimen
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization, and must not be breastfeeding and must agree to use contraceptive for duration of study.
* Participation in a clinical trial with an investigational therapy within 30 days prior to randomization
* Co-morbid disease or condition that would place the patient at undue risk and preclude safe use of TheraSphere treatment, in the Investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Mulcahy, MD, Principal Investigator — Northwestern University
Locations (131):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Fransico, Moffitt Hospital, San Francisco, California
  - University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado
  - Christiana Care Hospital, Newark, Delaware
  - Lynn Clinical Research Center, Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Miami Miller School of Medicine, Florida, Miami, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle Clinic, Urbana, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State Harper Hospita Karmanos Cancer Institute, Farmington Hills, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Aria Health, Trevose, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - St. Marks Hospital, Salt Lake City, Utah
  - Sentara Norfolk General, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Gundersen Medical Foundation, La Crosse, Wisconsin
  - Medical College of Wisconsin/Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Aurora Research Institute, Wauwatosa, Wisconsin
- Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - Onze-Lieve-Vrouwziekenuis VZW Campus Aalst, Aalst
  - AZ - Sint Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - QEII Health Services Center, Halifax Infirmary Site, Halifax, Nova Scotia
  - London Regional Cancer program, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network , Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Center - Glen Site, Montreal, Quebec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (2):
  - Hong Kong Sanatorium Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- France (14):
  - CHRU Montpellier - Hopital St Eloi, Montpellier, Cedex 5
  - CUH d'Angers, Angers, Cedex 9
  - CHU Toulouse, Hôpital Rangueil, Toulouse, Cedex 9
  - Institut Bergognié, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier Lyon-Sud, Lyon
  - Hôpital La Timone, Marseille
  - CHU Nantes-Hôtel Dieu, Nantes
  - CHU de Nice,, Hopital Archet 2 - Service d'Imagerie Médicale niveau -2, Nice
  - CHU Bordeaux, Pessac
  - Hôpital La Milétrie, CHU Poitiers, hépato gastroenterologie, Poitiers
  - Centre Eugene Marquis, Rennes
- Germany (8):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - SLK Kliniken, Heilbronn GmbH, Heilbronn
  - Universitätsklinikum des Saarlandes, Homburg
  - University Hospital of Leipzig, Leipzig
  - Universitaetsklinikum Marburg Klinik für Dermatologie und Allergologie, Marburg
  - Eberhard-Karls-University Tübingen, Tübingen
- Azienda Ospedaliera-Universitaria, Policlinico Sant'Orsola Malpighi, Bologna, Italy
- Poland (8):
  - Białostockie Centrum Onkologii, Bialystok
  - Centrum Onkologii - Instytut, im. Marii Skłodowskiej-Curie, Gliwice
  - Regionalny Szpital Specjalistyczny im. Dr Władysława Biegańskiego, Grudziądz
  - Oddział Onkologii Klinicznej; Centrum Onkologii Ziemi Lubelskiej im. Św.Jana z Dukli., Lublin
  - Szpital Kliniczny im. Heliodora Święcickiego, Poznan
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Centrum Onkologii - Instytut, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- National University Hospital, Singapore, Singapore
- South Korea (5):
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - St. Mary's Hospital, Seoul
- Spain (18):
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario del Henares, Coslada
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Avenida de Roma, s/n, Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Central de Asturias, Oviedo
  - Parc Taulí Sabadell Hospital Universitari, Sabadell
  - Hospital Universitari i Politècnic La Fe, Valencia
  - HCU Lozano Blesa, Planta 11-Oncología-Secretaría, Zaragoza
- United Kingdom (27):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital Bath NHS Trust, Bath
  - The Clatterbrdige Cancer Centre NHSF Trust, Bebington
  - Queen Elizabeth Hospital Cancer Centre, Birmingham
  - The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust - Royal Bournemouth Hospital, Bournemouth
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology and Oncology Centre, Bristol
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson Cancer Centre and University of Glasgow, Glasgow
  - University of Glasgow, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Calderdale and Huddersfield NHS Foundation Trust - Huddersfield Royal Infirmary, Huddersfield
  - Leeds Hospitals NHS Trust, Leeds
  - UCLH, University College London Hospitals, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospital NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust Churchill Hospital, Oxford
  - Barking, Havering and Redbridge University Hospitals NHS Trust - Queen's Hospital, Romford
  - Western Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Great Western Hospitals NHS Foundation Trust - The Great Western Hospital, Swindon
  - Taunton and Somerset NHS Foundation Trust - Musgrove Park Hospital, Taunton
  - Walsall Healthcare NHS Trust - Manor Hospital, Walsall
  - The Royal Wolverhampton NHS Trust - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Salem R, Garin E, Boucher E, Fowers K, Lam M, Padia S, Harris W. Optimal patient selection for yttrium-90 glass plus chemotherapy in the treatment of colorectal liver metastases: additional quality of life, efficacy, and safety analyses from the EPOCH study. Oncologist. 2024 Aug 5;29(8):681-689. doi: 10.1093/oncolo/oyae128. PMID 38985849
- [Derived] Mulcahy MF, Mahvash A, Pracht M, Montazeri AH, Bandula S, Martin RCG 2nd, Herrmann K, Brown E, Zuckerman D, Wilson G, Kim TY, Weaver A, Ross P, Harris WP, Graham J, Mills J, Yubero Esteban A, Johnson MS, Sofocleous CT, Padia SA, Lewandowski RJ, Garin E, Sinclair P, Salem R; EPOCH Investigators. Radioembolization With Chemotherapy for Colorectal Liver Metastases: A Randomized, Open-Label, International, Multicenter, Phase III Trial. J Clin Oncol. 2021 Dec 10;39(35):3897-3907. doi: 10.1200/JCO.21.01839. Epub 2021 Sep 20. PMID 34541864
- [Derived] Chauhan N, Mulcahy MF, Salem R, Benson Iii AB, Boucher E, Bukovcan J, Cosgrove D, Laframboise C, Lewandowski RJ, Master F, El-Rayes B, Strosberg JR, Sze DY, Sharma RA. TheraSphere Yttrium-90 Glass Microspheres Combined With Chemotherapy Versus Chemotherapy Alone in Second-Line Treatment of Patients With Metastatic Colorectal Carcinoma of the Liver: Protocol for the EPOCH Phase 3 Randomized Clinical Trial. JMIR Res Protoc. 2019 Jan 17;8(1):e11545. doi: 10.2196/11545. PMID 30664496

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 215 | 213
Completed | 169 | 153
Not Completed | 46 | 60
Not completed — Administrative Reasons | 2 | 1
Not completed — Withdrawal by Subject | 21 | 32
Not completed — Discontinuation by Investigator or Sponsor for any reason | 22 | 24
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 215 | 213 | 428
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 132 | 258
  >=65 years | 89 | 81 | 170
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 75 | 155
  Male | 135 | 138 | 273
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 164 | 169 | 333
  Black or African American | 9 | 8 | 17
  Asian | 25 | 17 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 1 | 1 | 2
  Missing | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  Singapore | 5 | 2 | 7
  United States | 54 | 50 | 104
  United Kingdom | 52 | 75 | 127
  Spain | 22 | 17 | 39
  Canada | 9 | 6 | 15
  Austria | 0 | 2 | 2
  South Korea | 13 | 9 | 22
  Belgium | 4 | 0 | 4
  Hong Kong | 3 | 1 | 4
  Poland | 28 | 28 | 56
  France | 15 | 18 | 33
  Germany | 10 | 5 | 15
Baseline Characteristics [Count of Participants; unit: Participants] — Patients with an ECOG Performance Status of 0 may have better overall response to treatment and fewer adverse events than those with an ECOG of 1 although both populations are considered to be relatively good candidates for this type of study Population: Three patients without baseline ECOG status are excluded from this analysis
  Participants
    number analyzed (Participants) | 214 | 211 | 425
    ECOG 0 at baseline | 119 | 133 | 252
    ECOG 1 at baseline | 95 | 78 | 173
KRAS status [Count of Participants; unit: Participants] — KRAS status: patients with a mutated KRAS may respond differently to targeted agents than those with KRAS wildtype which could lead to poorer response outcomes.
  Participants
    KRAS mutant | 100 | 101 | 201
    KRAS wildtype | 115 | 112 | 227
Unilobar vs Bilobar disease at baseline [Count of Participants; unit: Participants] — Metastatic disease from colorectal cancer to both lobes of the liver (bilobar) may be associated with poorer prognosis than patients presenting with disease to only one lobe (and potentially lower tumor burden).
  Participants
    unilobar | 39 | 40 | 79
    bilobar | 176 | 173 | 349

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free survival by blinded independent central review per RECIST 1.1
Time Frame: From date of randomization until the date of first documented progression, as defined by RECIST 1:1 or date of death from any cause, whichever comes first, assessed up to a minimum of 1 year follow up or until study completion
Population: Outcome measurement includes data from all subjects in the ITT.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 215 | 213
Months | 8.0 [7.2 to 9.2] | 7.2 [5.7 to 7.6]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Analysis performed using a log-rank test; Test type: Superiority; p = 0.0013, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.54 to 0.88]

2. Primary Outcome: Hepatic Progression-Free Survival (HPFS)
Description: Hepatic Progression Free Survival (HPFS) by blinded independant central review per RECIST 1.1
Time Frame: Time from randomization until hepatic PD by BICR per RECIST 1.1 or death, whichever occurs first, assessed up to a minimum of 1 year follow up or study completion.
Population: Outcome measurement includes data from all subjects in the ITT.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 215 | 213
Months | 9.1 [7.8 to 9.7] | 7.2 [5.7 to 7.6]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Analysis performed using a log-rank test; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.46 to 0.77]

3. Secondary Outcome: Overall Survival
Description: Time from randomization until date of death due to any cause as reported by study site.
Time Frame: Time from date of randomization until date of death due to any cause; patients remaining on study post progression were followed until study completion; duration of follow up could be a few months to several years depending on when event was met.
Population: ITT: all randomized patients with patient analyzed according to the treatment group to which they were randomized
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 215 | 213
Months | 14 [11.8 to 15.5] | 14.4 [12.8 to 16.4]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected until progression of disease or 30 days following discontinuation date of study therapy (chemo or TheraSphere), whichever comes first, on average up to 6 months depending on number of chemo cycles. After this only AEs, SAEs related to TheraSphere were collected through study completion, on average up to one year post treatment. All-cause mortality was collected through study completion, on average up to two years after first study treatment.
Description: Adverse events presented here are based on the Safety Population: all randomized patients who received at least 1 administration of TheraSphere or chemotherapy with patients analyzed according to the treatment they received (TheraSphere +Chemo=187 and Chemo only=207) with the exception of All Cause Mortality. For All Cause Mortality the Intent to Treat Population was utilized (TheraSphere + Chemo= 215 and Chemo only =213).
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 182/215 | 165/213
Serious Adverse Events (participants affected / at risk) | 95/187 | 47/207
Other Adverse Events (participants affected / at risk) | 186/187 | 196/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=187) | Control Group (N=207)
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 (9) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 3 (5)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 4 (4)
Ascites (Gastrointestinal disorders) | 11 (15) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 4 (4) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (8) | 2 (3)
General physical health deterioration (General disorders) | 2 (2) | 3 (3)
Disease progression (General disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 4 (4) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (3)
Device related sepsis (Infections and infestations) | 1 (1) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (2)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fungal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster opthalmic (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation hepatitis (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Influenza B virus test positive (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
death (General disorders) | 1 (1) | 0 (0) — Death was of unknown cause, there is no known specific adverse event term associated with this death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=187) | Control Group (N=207)
Neutropenia (Blood and lymphatic system disorders) | 64 (172) | 50 (99)
Thrombocytopenia (Blood and lymphatic system disorders) | 38 (89) | 19 (37)
Anaemia (Blood and lymphatic system disorders) | 26 (39) | 11 (16)
Leukopenia (Blood and lymphatic system disorders) | 19 (29) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 8 (12) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 4 (7)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 4 (7) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac disorders (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Artial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (5) | 4 (5)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 4 (4)
Dry eye (Eye disorders) | 2 (2) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 3 (3)
Vision blurred (Eye disorders) | 2 (2) | 2 (2)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 90 (164) | 90 (176)
Diarrhoea (Gastrointestinal disorders) | 62 (127) | 102 (225)
Constipation (Gastrointestinal disorders) | 63 (86) | 49 (76)
Abdominal pain (Gastrointestinal disorders) | 68 (117) | 41 (48)
Vomiting (Gastrointestinal disorders) | 48 (85) | 35 (52)
Stomatitis (Gastrointestinal disorders) | 24 (42) | 33 (72)
Abdominal pain upper (Gastrointestinal disorders) | 26 (31) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 24 (29) | 11 (18)
Ascites (Gastrointestinal disorders) | 27 (42) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 14 (17) | 6 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 7 (8) | 9 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (9) | 6 (7)
Proctalgia (Gastrointestinal disorders) | 8 (9) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 5 (5)
Flatulence (Gastrointestinal disorders) | 5 (5) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Toothache (Gastrointestinal disorders) | 5 (5) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 6 (6) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 3 (3) | 2 (3)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (3) | 3 (4)
Gastritis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (4) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 2 (3) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 4 (4) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Anal inflammation (Gastrointestinal disorders) | 3 (7) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (2) | 2 (2)
Chelitis (Gastrointestinal disorders) | 0 (0) | 2 (6)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Painful defaecation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 91 (206) | 94 (210)
Mucosal inflammation (General disorders) | 20 (40) | 41 (86)
Pyrexia (Gastrointestinal disorders) | 40 (56) | 21 (26)
Asthenia (Gastrointestinal disorders) | 30 (79) | 18 (53)
Oedema peripheral (General disorders) | 19 (24) | 10 (16)
Chills (General disorders) | 9 (12) | 8 (9)
Non-cardiac chest pain (General disorders) | 7 (8) | 2 (3)
Pain (General disorders) | 4 (4) | 5 (7)
Catheter site pain (General disorders) | 5 (5) | 3 (4)
General physical health deterioration (General disorders) | 2 (2) | 4 (4)
Oedema (General disorders) | 5 (7) | 1 (1)
Chest pain (General disorders) | 2 (2) | 3 (4)
Disease progression (General disorders) | 3 (3) | 2 (2)
Catheter site erythema (General disorders) | 2 (2) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 3 (3)
Device component issue (General disorders) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 3 (3)
Thrombosis in device (General disorders) | 1 (1) | 2 (2)
Catheter site haematoma (General disorders) | 2 (2) | 0 (0)
Catheter site inflammation (General disorders) | 2 (2) | 0 (0)
Catheter site rash (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Secretion discharge (General disorders) | 1 (1) | 1 (1)
Temperature intolerance (General disorders) | 1 (2) | 1 (1)
Vessel puncture site pain (General disorders) | 2 (2) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Obstruction (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 6 (8) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 3 (3) | 3 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 (8) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 5 (5) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Portal hypertension (Hepatobiliary disorders) | 3 (3) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (3) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 7 (7)
Hypersensitivity (Immune system disorders) | 3 (5) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 13 (14)
Urinary tract infection (Infections and infestations) | 15 (17) | 8 (12)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (7)
Lower respiratory tract infection (Infections and infestations) | 5 (6) | 7 (7)
Oral candidiasis (Infections and infestations) | 6 (7) | 6 (8)
Rash pustular (Infections and infestations) | 4 (4) | 6 (15)
Sepsis (Infections and infestations) | 6 (6) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4)
Catheter site infection (Infections and infestations) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3)
Tooth abscess (Infections and infestations) | 1 (1) | 4 (5)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 4 (4)
Candidiasis (Infections and infestations) | 3 (4) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 2 (3) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (3)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (3)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Ependymitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (2)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster opthalmic (Infections and infestations) | 0 (0) | 1 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (2)
Joint abscess (Infections and infestations) | 1 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (3)
Omphalitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Propionibacterium infection (Infections and infestations) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation hepatitis (Injury, poisoning and procedural complications) | 8 (9) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Infusion relation reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 51 (67) | 47 (63)
alopecia (Skin and subcutaneous tissue disorders) | 23 (27) | 43 (47)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 26 (45)
cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 22 (23)
neuropathy peripheral (Nervous system disorders) | 25 (49) | 35 (57)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 21 (27)
hypertension (Vascular disorders) | 20 (24) | 18 (43)
anemia (Blood and lymphatic system disorders) | 26 (39) | 11 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (25) | 17 (45)
Neutrophil count decreased (Investigations) | 16 (23) | 20 (20)
headache (Nervous system disorders) | 15 (15) | 19 (35)
insomnia (Psychiatric disorders) | 17 (26) | 15 (17)
rash (Skin and subcutaneous tissue disorders) | 21 (36) | 10 (18)
back pain (Musculoskeletal and connective tissue disorders) | 17 (19) | 14 (19)
Blood alkaline phosphatase increased (Investigations) | 21 (27) | 8 (12)
weight decreased (Investigations) | 13 (16) | 15 (20)
dizziness (Nervous system disorders) | 19 (21) | 8 (9)
Dysgeusia (Nervous system disorders) | 10 (12) | 15 (16)
Platelet count decreased (Investigations) | 15 (23) | 9 (14)
hypokalemia (Metabolism and nutrition disorders) | 14 (25) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 16 (27) | 4 (5)
abdominal distention (Gastrointestinal disorders) | 14 (17) | 6 (6)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 9 (10)
Paraesthesia (Nervous system disorders) | 7 (14) | 12 (25)
Blood bilirubin increased (Investigations) | 18 (27) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (20) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (12) | 6 (15)
muscle spasm (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 (15) | 0 (0)
Lymphocyte count decreased (Investigations) | 10 (12) | 2 (4)

LIMITATIONS AND CAVEATS:
For the event of death noted as "other" this is how it was captured in our database due to fact that it was a death "unknown cause" and there is no related SAE. It is captured as an event under All Cause Mortality table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT01483027/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT01483027/SAP_001.pdf